CLINICAL TRIAL: NCT04611919
Title: Prevalence of Sexually Transmitted Infections (STIs) at Entry Into Prison in Reunion
Brief Title: Prevalence of Sexually Transmitted Infections (STIs) Into Prison in Reunion
Acronym: PRECARIST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/11
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the beginning of the 2000s, there has been a steady increase in the incidence of STIs in France. In Reunion, the few figures available seem to show the same phenomenon, especially for syphilis. The unfavorable socio-economic context, which is characterized by high levels of precariousness, significant population exchanges (immigration, travel) with neighboring countries, behaviors around sexuality or screening for STIs different from those observed in mainland France are all factors testify to the singularity of the Reunion island in relation to the metropolitan France with regard to the risk factors of STIs.

STI management has become a priority in public health; in particular, the 2010-2014 HIV and STI control plan emphasized the need for their surveillance and screening. These are often asymptomatic infections that can cause serious complications if they are not treated (infertility, ectopic pregnancies, maternal-fetal infections, ...). Screening them in at-risk populations is therefore essential to reduce their prevalence.

The prison population is a vulnerable population, possibly exposed during the incarceration but also upstream of it (generally low levels of education, over-represented disadvantaged social categories, low access and use of care, high prevalence of risky behaviors). ). Some prevalence studies of STIs in these populations have been carried out in metropolitan France, indicating a prevalence higher than that observed in the general population. There is little data on the subject for the prison population in Réunion; Given the local specificities, it seems necessary to improve the epidemiological knowledge of STIs in this prison population in Réunion, in order to be able to adapt the prevention and care measures, the conditions of detention presenting potentially aggravating situations (promiscuity, confinement). , hygienic conditions, ...).

ELIGIBILITY:
Inclusion Criteria:

* imprisoned at Domenjod prison between 01/02/2018 and on 04/30/2019
* able to answer a questionnaire,
* domiciled in Réunion at the time of incarceration,
* incarceration medical examination carried out within 7 days incarceration,

Exclusion Criteria:

* incarcerated by transfer from another penal institution
* having had antibiotic therapy in the 3 months before the inclusion consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Screening will be offered to all adults entering prison at Domenjod prison (Reunion Island) between 01/02/2018 and 30/04/2019.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sexually Transmitted Infection with Chlamydia trachomatis, Neisseria gonorrheae and Mycoplasma genitalium | Day 1
  Proportion of people with a positive triplex Polymerase Chain Reaction result of detection of Chlamydia trachomatis, Neisseria gonorrheae and/or Mycoplasma genitalium on samples.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre MOITON, MD, Principal Investigator — CHU de La Réunion
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, Saint-Denis, Reunion